CLINICAL TRIAL: NCT00994760
Title: A Prospective Non-interventional/Observational Patient Cohort Study on the Efficacy of Intranasal Fentanyl Spray for the Treatment of Breakthrough Pain in Cancer Patients.
Brief Title: Efficacy and Tolerability of Intranasal Fentanyl Spray for the Treatment of Breakthrough Pain in Cancer Patients Older Than 18 Years
Acronym: GENISIS
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: FT-1301-401-DE
Record Dates: First submitted 2009-10-05; First posted 2009-10-14 (Estimated); Results first posted 2012-09-27 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-08

CONDITIONS: Breakthrough Pain; Cancer
Keywords: intranasal fentanyl spray
MeSH Terms: conditions — Breakthrough Pain; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GENISIS
  Interventions: Drug: Instanyl (Intranasal Fentanyl)

INTERVENTIONS:
Drug: Instanyl (Intranasal Fentanyl) — This was an observational study. Therefore, the physician decided about dosage according to individual needs.

SUMMARY:
The aim of the study was to evaluate the safety and efficacy of intranasal fentanyl spray in cancer patients over four weeks, especially during cancer-related breakthrough pain (BTP) attacks. The fentanyl spray was applied into the nose by a metered-spray device. The study was to provide further data on pharmacoeconomic efficiency of intranasal fentanyl spray.

ELIGIBILITY:
Inclusion criteria:

* decision to start treatment with intranasal fentanyl spray
* written informed consent

Exclusion criteria:

* criteria as defined in the Summary of Product Characteristics (Fachinformation Chapter 4.3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Thomas D. Bethke, PhD; MD, Study Director — Nycomed Deutschland GmbH, 78467 Konstanz, Germany
Locations (128):
- Germany (128):
  - Nycomed Deutschland GmbH, Aachen
  - Nycomed Deutschland GmbH, Adendorf
  - Nycomed Deutschland GmbH, Aichach
  - Nycomed Deutschland GmbH, Albstadt
  - Nycomed Deutschland GmbH, Albstadt-Ebingen
  - Nycomed Deutschland GmbH, Altenkirchen
  - Nycomed Deutschland GmbH, Aschaffenburg
  - Nycomed Deutschland GmbH, Aschersleben
  - Nycomed Deutschland GmbH, Augsburg
  - Nycomed Deutschland GmbH, Backnang
  - Nycomed Deutschland GmbH, Bad Bevensen
  - Nycomed Deutschland GmbH, Bad Dürkheim
  - Nycomed Deutschland GmbH, Bad Liebenstein
  - Nycomed Deutschland GmbH, Bad Pyrmont
  - Nycomed Deutschland GmbH, Bad Schwalbach
  - Nycomed Deutschland GmbH, Badel
  - Nycomed Deutschland GmbH, Bademühlen
  - Nycomed Deutschland GmbH, Bautzen
  - Nycomed Deutschland GmbH, Berlin
  - Nycomed Deutschland GmbH, Bochum
  - Nycomed Deutschland GmbH, Bonn
  - Nycomed Deutschland GmbH, Böblingen
  - Nycomed Deutschland GmbH, Brandenburg/Havel
  - Nycomed Deutschland GmbH, Braunschweig
  - Nycomed Deutschland GmbH, Bremen
  - Nycomed Deutschland GmbH, Brühl
  - Nycomed Deutschland GmbH, Burg
  - Nycomed Deutschland GmbH, Burg/Fehmarn
  - Nycomed Deutschland GmbH, Burscheid
  - Nycomed Deutschland GmbH, Butzbach
  - Nycomed Deutschland GmbH, Coburg
  - Nycomed Deutschland GmbH, Cochem
  - Nycomed Deutschland GmbH, Cologne
  - Nycomed Deutschland GmbH, Cottbus
  - Nycomed Deutschland GmbH, Cuxhaven
  - Nycomed Deutschland GmbH, Dessau
  - Nycomed Deutschland GmbH, Dresden
  - Nycomed Deutschland GmbH, Duisburg
  - Nycomed Deutschland GmbH, Düsseldorf
  - Nycomed Deutschland GmbH, Essen
  - Nycomed Deutschland GmbH, Etzenricht
  - Nycomed Deutschland GmbH, Fehmarn
  - Nycomed Deutschland GmbH, Frankfurt
  - Nycomed Deutschland GmbH, Freiburg im Breisgau
  - Nycomed Deutschland GmbH, Friedberg
  - Nycomed Deutschland GmbH, Geesthacht
  - Nycomed Deutschland GmbH, Göppingen
  - Nycomed Deutschland GmbH, Görlitz
  - Nycomed Deutschland GmbH, Großheirath-Rossach
  - Nycomed Deutschland GmbH, Gütersloh
  - Nycomed Deutschland GmbH, Hachenburg
  - Nycomed Deutschland GmbH, Hainburg
  - Nycomed Deutschland GmbH, Halle
  - Nycomed Deutschland GmbH, Hamburg
  - Nycomed Deutschland GmbH, Hamelin
  - Nycomed Deutschland GmbH, Hanover
  - Nycomed Deutschland GmbH, Heidelberg
  - Nycomed Deutschland GmbH, Hellenthal
  - Nycomed Deutschland GmbH, Herne
  - Nycomed Deutschland GmbH, Herzlake
  - Nycomed Deutschland GmbH, Hohberg
  - Nycomed Deutschland GmbH, Hohberg-Hofweiler
  - Nycomed Deutschland GmbH, Holzminden
  - Nycomed Deutschland GmbH, Husum
  - Nycomed Deutschland GmbH, Iserlohn
  - Nycomed Deutschland GmbH, Itzehoe
  - Nycomed Deutschland GmbH, Jerichow
  - Nycomed Deutschland GmbH, Kaiserslautern
  - Nycomed Deutschland GmbH, Karlsbad
  - Nycomed Deutschland GmbH, Katzhütte
  - Nycomed Deutschland GmbH, Kevelaar
  - Nycomed Deutschland GmbH, Kiel
  - Nycomed Deutschland GmbH, Kirchberg
  - Nycomed Deutschland GmbH, Koblenz
  - Nycomed Deutschland GmbH, Köthen
  - Nycomed Deutschland GmbH, Krefeld
  - Nycomed Deutschland GmbH, Laatzen
  - Nycomed Deutschland GmbH, Lage/Lippe
  - Nycomed Deutschland GmbH, Landshut
  - Nycomed Deutschland GmbH, Leipzig
  - Nycomed Deutschland GmbH, Leverkusen
  - Nycomed Deutschland GmbH, Ludwigshafen
  - Nycomed Deutschland GmbH, Magdeburg
  - Nycomed Deutschland GmbH, Mainz
  - Nycomed Deutschland GmbH, Mannheim
  - Nycomed Deutschland GmbH, Mayen
  - Nycomed Deutschland GmbH, Meinersen
  - Nycomed Deutschland GmbH, München
  - Nycomed Deutschland GmbH, Nastätten
  - Nycomed Deutschland GmbH, Naumburg
  - Nycomed Deutschland GmbH, Neubrandenburg
  - Nycomed Deutschland GmbH, Neuss
  - Nycomed Deutschland GmbH, Neustadt
  - Nycomed Deutschland GmbH, Nordhorn
  - Nycomed Deutschland GmbH, Olpe
  - Nycomed Deutschland GmbH, Osloß
  - Nycomed Deutschland GmbH, Osnabrück
  - Nycomed Deutschland GmbH, Pforzheim
  - Nycomed Deutschland GmbH, Plate
  - Nycomed Deutschland GmbH, Plüderhausen
  - Nycomed Deutschland GmbH, Potsdam
  - Nycomed Deutschland GmbH, Potsdam-Babelsberg
  - Nycomed Deutschland GmbH, Pulheim-Stommeln
  - Nycomed Deutschland GmbH, Quedlinburg
  - Nycomed Deutschland GmbH, Rheine
  - Nycomed Deutschland GmbH, Rosenfeld
  - Nycomed Deutschland GmbH, Rostock
  - Nycomed Deutschland GmbH, Sangerhausen
  - Nycomed Deutschland GmbH, Sankt Michaelisdonn
  - Nycomed Deutschland GmbH, Schleswig
  - Nycomed Deutschland GmbH, Siegen
  - Nycomed Deutschland GmbH, Solingen
  - Nycomed Deutschland GmbH, Stendal
  - Nycomed Deutschland GmbH, Stuttgart
  - Nycomed Deutschland GmbH, Tangermünde
  - Nycomed Deutschland GmbH, Ulm
  - Nycomed Deutschland GmbH, Varel
  - Nycomed Deutschland GmbH, Velbert
  - Nycomed Deutschland GmbH, Villingen-Schwenningen
  - Nycomed Deutschland GmbH, Wedel
  - Nycomed Deutschland GmbH, Weinsberg
  - Nycomed Deutschland GmbH, Werdau
  - Nycomed Deutschland GmbH, Wesendorf
  - Nycomed Deutschland GmbH, Westhausen
  - Nycomed Deutschland GmbH, Wiesbaden
  - Nycomed Deutschland GmbH, Wilster
  - Nycomed Deutschland GmbH, Zwickau
  - Nycomed Deutschland GmbH, Zwönitz

RESULTS

PARTICIPANT FLOW:
Groups:
- GENISIS: Intranasal Fentanyl Spray
Period: Overall Study
Arm/Group | GENISIS
Started | 131
Completed | 107
Not Completed | 24

BASELINE CHARACTERISTICS:
Arm/Group | GENISIS
Number analyzed (Participants) | 131
Age Continuous [Mean (Standard Deviation); unit: years] — Number of valid cases = 130. Number of valid cases = patients with data available.
  years | 62.1 (12.1)
Sex/Gender, Customized [Number; unit: participants]
  Female | 60
  Male | 67
  Missing | 4
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kgˆm2] — Number of valid cases = 126. Number of valid cases = patients with data available.
  kgˆm2 | 23.2 (4.4)
Tumor diagnosis (malignant neop-lasms ICD10) [Number; unit: percentage of participants]
  Pain not caused by tumor | 2.3
  C00-C14 lip, oral cavity and pharynx | 6.1
  C15-C26 digestive organs | 26.0
  C30-C39 respiratory and intrathoracic organs | 16.0
  C40-C41 bone and articular cartilage | 0.8
  C43-C44 Melanoma and other skin | 0.8
  C50-C50 Mamma | 20.6
  C51-C58 female genital organs | 3.1
  C60-C63 male genital organs | 13.0
  C64-C68 urinary tract | 5.3
  C73-C75 thyroid and other endocrine glands | 0.8
  C76-C80 ill-defined, secondary + unspecified sites | 0.8
  C81-C96 lymphoid, hematopoietic and related tissue | 0.8
  Missing | 3.8
Karnofsky-index [Mean (Standard Deviation); unit: scores] — score 0= worst (death) , 100= best (no limitation in health)
  Number of valid cases = 125. Number of valid cases = patients with data available.
  scores | 58.6 (21.6)
American Society of Anesthesiologists (ASA)-physical state (2-5) [Number; unit: participants] — ASA = physical status.
  * state 2: patient with slight generalized disease
  * state 3: patient with severe generalized disease
  * state 4: life threatening generalized disease
  * state 5: moribund patient, unlikly to survive without operation
  participants
    ASA 2 | 22
    ASA 3 | 40
    ASA 4 | 59
    ASA 5 | 5
    Missing | 5
ECOG (Eastern Cooperative Oncology Group) performance status (0-4) [Number; unit: participants] — ECOG 0 (fully active) ECOG 1 (restricted in strenuous activity, ambulatory) ECOG 2 (ambulatory, up and about more than 50% of waking hours ECOG 3 (limited selfcare, confined to bed > 50% of waking hours ECOG 4 (completely disabled, no selfcare)
  participants
    ECOG 0 | 2
    ECOG 1 | 33
    ECOG 2 | 40
    ECOG 3 | 36
    ECOG 4 | 14
    Missing | 6
Reason for the use of Instanyl [Number; unit: participants] — (multiple reasons possible)
  participants
    No previous BTP medication | 86
    Previous BTP medic./Insufficient efficacy | 32
    Previous BTP medic./Insufficient speed of action | 32
    Previous BTP medic./Insufficient handling | 12
    Previous BTP medic./Insufficient tolerability | 6
    Previous BTP medic./Other reasons | 7

OUTCOME MEASURES:

1. Primary Outcome: Dose of Instanyl
Description: Initially prescribed dose/ most efficient single dose of Instanyl at study end
Time Frame: during therapy with Instanyl (planned: 28 days)
Population: Patients included and treated (without imputation of missing values), intention to treat.
  All patients included
Measure: Number; unit: participants
Arm/Group | Study Start | Study End
Number analyzed (Participants) | 131 | 116
participants
  50 µg | 75 | 30
  100 µg | 50 | 69
  200 µg | 5 | 15
  400 µg | 0 | 1
  Missing | 1 | 1

2. Primary Outcome: Physician: Degree of Maximum Pain Intensity During the Last Days/ Since the Last Examination
Description: Scale: 0=no, 1=mild, 2=moderate, 3=strong, 4=very strong, 5=extreme
Time Frame: before and after therapy with Instanyl (first/last visit)
Population: All patients included and treated, intention to treat, missing values not imputed.
  All patients with valid values ('as observed'). N= number of valid cases.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Initial Visit | Last Visit
Number analyzed (Participants) | 131 | 116
units on a scale
  Persistent pain (IV: N= 126, LV: N= 116) | 2.3 (1.1) | 1.6 (0.9)
  Breakthrough pain (IV: N= 126, LV: N= 115) | 3.5 (0.9) | 1.8 (1.2)

3. Secondary Outcome: Physician: Degree of Relief of Breakthrough Pain Achieved by Instanyl at Study End
Description: 0=no reduction, 1=slight, 2=medium, 3=strong, 4=very strong, 5=complete
Time Frame: after therapy with Instanyl (planned: 4 weeks)
Population: Patients included and treated with valid data (without imputation of missing values), intention to treat.
  All patients with valid values at last visit. N= number of valid cases (=114). From the 116 participants analyzed, only 114 participants had valid values at the last visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Last Visit
Number analyzed (Participants) | 116
units on a scale | 3.4 (1.0)

4. Primary Outcome: Physician: Assessment of Breakthrough Pain Therapy (Initial Visit: Previous/Last Visit: Instanyl)
Description: Scale: 1=very good, 2=good, 3=satisfactory, 4=poor, 5=very poor, 6=insufficient
Time Frame: before and after therapy with Instanyl (first/last visit)
Population: All patients included and treated, intention to treat, missing values not imputed.
  All patients with valid values ('as observed')= N.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | First Visit (FV): Patients With Previous BTP- Medication Only | Last Visit (LV)
Number analyzed (Participants) | 45 | 116
units on a scale
  speed of action (FV: N= 45, LV: N= 114) | 4.0 (1.3) | 1.7 (0.8)
  strength of action (FV: N= 45, LV: N= 115) | 4.0 (1.3) | 1.8 (0.9)
  tolerability (FV: N= 44, LV: N= 113) | 3.0 (1.4) | 1.7 (0.6)
  safety (FV: N= 45, LV: N= 114) | 2.9 (1.2) | 1.7 (0.6)
  handling (FV: N= 45, LV: N= 115) | 3.4 (1.4) | 2.1 (1.2)
  patient satisfaction (FV: N= 45, LV: N= 116) | 4.2 (1.3) | 1.9 (1.1)

5. Primary Outcome: Physician: To What Extent Did Your Expectations in Instanyl Have Met? (Last Visit)
Description: 5=completely, 4=for the most part, 3=partially, 2= more or less, 1=rather not, 0=not at all
Time Frame: after therapy with Instanyl (planned: 4 weeks)
Population: Patients included and treated with valid data (without imputation of missing values), intention to treat.
  All patients with valid values at last visit. N= number of valid cases (=110). From the 116 participants analyzed, only 110 participants had valid values at the last visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Physician Last Visit (LV)
Number analyzed (Participants) | 116
units on a scale | 4.4 (0.7)

6. Primary Outcome: Physician: To What Extent Changes Have Occurred Induced by the Treatment of Breakthrough Pain With Instanyl With Respect to ... (at Last Visit)
Description: Scale: -3= very much improved, -2= much improved, -1= improved, 0= comparable, 1= worsened, 2= much worsened ,3= very much worsened
Time Frame: after therapy with Instanyl (at last visit)
Population: All patients included and treated, intention to treat, missing values not imputed.
  All patients with valid values ('as observed'). N=number of valid cases.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GENISIS
Number analyzed (Participants) | 116
units on a scale
  Nursing and support efforts (N= 113) | -1.2 (1.0)
  Autonomy of the patient (N= 113) | -1.5 (0.9)
  Pain-related impairment in everyday life (N= 113) | -1.6 (0.9)
  Quality of patient's life (N= 112) | -1.5 (0.9)
  Extent of use of other medical services (N= 112) | -1.1 (1.0)

7. Primary Outcome: Physician: What is the Current Treatment Needs of Your Patient Regarding ...
Description: Scale: 0=no, 1=low, 2=medium, 3=high
Time Frame: before and after therapy with Instanyl (first/last visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Initial Visit (IV) | Last Visit (LV)
Number analyzed (Participants) | 131 | 116
units on a scale
  persistent pain (IV: N=131, LV: N=112) | 2.0 (0.8) | 1.3 (0.8)
  breakthrough pain (IV: N=130, LV: N=111) | 2.5 (0.6) | 1.2 (0.8)
  nausea (IV: N=130, LV: N=112) | 1.5 (0.8) | 0.9 (0.8)
  vomiting (IV: N=130, LV: N=112) | 1.2 (0.9) | 0.7 (0.7)
  dyspnoea (IV: N=130, LV: N=111) | 1.0 (0.9) | 0.7 (0.8)
  constipation (IV: N=129, LV: N=112) | 1.2 (0.9) | 0.8 (0.8)
  weakness (IV: N=129, LV: N=112) | 2.0 (0.8) | 1.4 (1.0)
  poor appetite (IV: N=131, LV: N=112) | 1.8 (0.9) | 1.4 (1.0)
  tiredness (IV: N=130, LV: N=112) | 1.8 (0.8) | 1.4 (0.9)
  efforts due to wounds/decubitus (N=130, N=112) | 1.0 (1.0) | 0.8 (0.9)
  need for assistance (IV: N=130, LV: N=111) | 1.8 (0.9) | 1.3 (0.9)
  depressiveness (IV: N=129, LV: N=111) | 1.6 (0.8) | 1.1 (0.8)
  anxiety (IV: N=130, LV: N=112) | 1.6 (0.8) | 1.1 (0.7)
  tension (IV: N=130, LV: N=112) | 1.6 (0.9) | 1.2 (0.8)
  disorientation, confusion (IV: N=130, LV: N=111) | 0.6 (0.8) | 0.5 (0.7)
  Problems with organization of care (N=129, N=112) | 1.1 (1.0) | 0.8 (0.8)
  Overburdening family/environment N=129, N=112 | 1.4 (1.0) | 1.0 (0.8)

8. Secondary Outcome: Patient: How Many Episodes of Pain You Experience on Average?
Time Frame: initial visit (before start of therapy with Instanyl)
Population: All patients included and treated who filled in the patient's documentation, intention to treat, missing values not imputed.
  All patients with valid values ('as observed'). N= number of valid cases (= 91). From the 95 participants analyzed, only 91 participants had valid values at the last visit.
Measure: Mean (Standard Deviation); unit: episodes per day
Arm/Group | First Visit
Number analyzed (Participants) | 95
episodes per day | 3.0 (2.2)

9. Secondary Outcome: Patient: Description of Pain at Initial Visit
Description: 0=no pain, 10= most intense pain imaginable
Time Frame: initial visit (before start of therapy with Instanyl)
Population: All patients included and treated who filled in the patient's documentation, intention to treat, missing values not imputed.
  All patients with valid values ('as observed') =N.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients at First Visit
Number analyzed (Participants) | 95
units on a scale
  Persistent pain in the last 24 hrs on average N=94 | 5.6 (2.3)
  Pain during the last pain attacks maximally N=93 | 8.3 (1.4)
  Pain intensity bearable N= 94 | 4.0 (1.5)

10. Secondary Outcome: Patient: How do You Feel Today?
Description: Scale: 1=very bad, 2=bad, 3=mediocre, 4=good, 5=very good
Time Frame: before and after therapy with Instanyl (first/last visit)
Population: All patients included and treated who filled in the patient's documentation, intention to treat, missing values not imputed.
  All patients with valid values ('as observed'). N= number of valid cases.
  * Initial Visit N=94
  * Last Visit N=83
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Initial Visit | Last Visit
Number analyzed (Participants) | 95 | 83
units on a scale | 2.2 (0.7) | 3.3 (0.8)

11. Secondary Outcome: Patient: To What Extent Your Present Condition is Affected by Your Pain Attacks?
Description: Scale: 0=not at all, 10=completely
Time Frame: before and after therapy with Instanyl (first/last visit)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Initial Visit | Last Visit
Number analyzed (Participants) | 95 | 83
units on a scale | 7.6 (1.7) | 3.8 (2.3)

12. Secondary Outcome: Patient: Modified Pain Disability Index (mPDI) - Sum - Score (Complete Questionnaires Only)
Description: Scale: 0=no impairment, 70=complete impairment
Time Frame: before and after therapy with Instanyl (first/last visit)
Population: All patients included and treated who filled in the patient's documentation, intention to treat, missing values not imputed.
  All patients with valid values ('as observed'). N= number of valid cases.
  * Initial Visit N=92
  * Last Visit N= 80
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Initial Visit | Last Visit
Number analyzed (Participants) | 95 | 83
units on a scale | 51.9 (11.4) | 29.1 (16.3)

13. Secondary Outcome: Patient: Quality-of-Life-Impairment by Pain =QLIP - Sum - Score (Complete Questionnaires Only)
Description: Scale: 0=complete impairment, 43=no impairment
Time Frame: before and after therapy with Instanyl (first/last visit)
Population: All patients included and treated who filled in the patient's documentation, intention to treat, missing values not imputed.
  All patients with valid values ('as observed'). N= number of valid cases.
  * Initial Visit N=93
  * Last Visit N=82
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Initial Visit | Last Visit
Number analyzed (Participants) | 95 | 83
units on a scale | 12.3 (6.6) | 24.7 (7.3)

14. Secondary Outcome: Patient: Quality-of-Life-Impairment by Pain =QLIP - Sum - Score (Complete Questionnaires Only) Conspicuous ≤20
Description: 0= conspicuous ≤20
  1= inconspicuous >20
Time Frame: before and after therapy with Instanyl (first/last visit)
Population: All patients included and treated who filled in the patient's documentation, intention to treat, missing values not imputed.
  All patients with valid values ('as observed'). N= number of valid cases.
Measure: Number; unit: participants
Arm/Group | Initial Visit | Last Visit
Number analyzed (Participants) | 95 | 83
participants
  QLIP - score (classified):QLIP conspicuous (≤20) | 80 | 21
  QLIP - score (classified):QLIP inconspicuous (>20) | 13 | 61
  Missing | 2 | 1

15. Secondary Outcome: Patient: Marburg Questionnaire on Habitual Health (MQHH): Sum - Score (Complete Questionnaires Only)
Description: Scale: 0=worst, 5=best
Time Frame: before and after therapy with Instanyl (first/last visit)
Population: All patients included and treated who filled in the patient's documentation, intention to treat, missing values not imputed.
  All patients with valid values ('as observed'). N= number of valid cases.
  * Initial Visit N=93
  * Last Visit N=81
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Initial Visit | Last Visit
Number analyzed (Participants) | 95 | 83
units on a scale | 1.2 (1.0) | 2.2 (1.2)

16. Secondary Outcome: Patient: Marburg Questionnaire on Habitual Health (MQHH): Sum - Score (Complete Questionnaires Only) Conspicuous <1.5
Description: conspicuous score <1.5 inconspicuous score ≥1.5
Time Frame: before and after therapy with Instanyl (first/last visit)
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Initial Visit | Last Visit
Number analyzed (Participants) | 95 | 83
participants
  MQHH - score (classified):conspicuous:score <1.5 | 62 | 24
  MQHH - score (classified):inconspicuous:score ≥1.5 | 31 | 57
  Missing | 2 | 2

17. Secondary Outcome: Patient: Degree of Relief of Breakthrough Pain Achieved by Instanyl at Study End
Description: 0=no reduction, 1=slight, 2=medium, 3=strong, 4=very strong, 5=complete
Time Frame: after therapy with Instanyl (planned: 4 weeks)
Population: Patients included and treated who filled in the patient's documentation with valid data (without imputation of missing values), intention to treat.
  All patients with valid values at last visit. N= number of valid cases (80). From the 83 participants analyzed, only 80 participants had valid values at the last visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients at Final Visit
Number analyzed (Participants) | 83
units on a scale | 3.4 (1.0)

18. Secondary Outcome: Patient: Assessment of Breakthrough Pain Therapy (Initial Visit: Previous/Last Visit: Instanyl)
Description: Scale: 1=very good, 2=good, 3=satisfactory, 4=poor, 5=very poor, 6=insufficient
Time Frame: before and after therapy with Instanyl (first/last visit)
Population: All patients included and treated who filled in the patient's documentation, intention to treat, missing values not imputed.
  All patients with valid values ('as observed').
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | First Visit (FV)(Patients With Previous BTP-medication Only) | Last Visit (LV)
Number analyzed (Participants) | 34 | 83
units on a scale
  speed of action (FV: N=33, LV: N=82) | 4.1 (1.1) | 2.0 (1.0)
  strength of action (FV: N=33, LV: N=82) | 3.9 (1.2) | 2.0 (1.1)
  tolerability (FV: N=33, LV: N=82) | 3.2 (1.1) | 2.0 (1.1)
  handling (FV: N=33, LV: N=80) | 3.4 (1.3) | 2.0 (1.0)
  total satisfaction (FV: N=NA, LV: N=82) | NA (NA) — no participants contributed data | 2.0 (1.1)

19. Secondary Outcome: Patient: To What Extent Did Your Expectations in Instanyl Have Met With Respect to ... (Last Visit)
Description: 5=completely, 4=for the most part, 3=partially, 2=more or less, 1=rather not, 0=not at all
Time Frame: after therapy with Instanyl (planned: 4 weeks)
Population: Patients included and treated who filled in the patient's documentation with valid data (without imputation of missing values), intention to treat.
  All patients with valid values at last visit. N= number of valid cases.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients at Final Visit
Number analyzed (Participants) | 83
units on a scale
  speed of action (N=79) | 4.2 (0.8)
  strength of action (N=80) | 4.2 (0.9)
  tolerability (N=78) | 4.3 (0.7)
  handling (N=79) | 4.2 (0.9)
  total satisfaction (N=80) | 4.2 (0.9)

20. Secondary Outcome: Patient: To What Extent Changes Have Occurred Induced by the Treatment of Breakthrough Pain With Instanyl With Respect to ...(at Last Visit)
Description: Scale: -3= very much improved, -2= much improved, -1= improved , 0= comparable, 1= worsened, 2= much worsened, 3= very much worsened
Time Frame: after therapy with Instanyl (at last visit)
Population: All patients included and treated who filled in the patient's documentation, intention to treat, missing values not imputed.
  All patients with valid values ('as observed'). N= number of valid cases (=81). From the 83 participants analyzed, only 81 participants had valid values at the last visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients at Final Visit
Number analyzed (Participants) | 83
units on a scale
  Nursing and support efforts (N= 81) | -1.0 (0.9)
  Autonomy of the patient (N= 81) | -1.4 (0.8)
  Pain-related impairment in everyday life (N= 81) | -1.3 (0.8)
  Quality of patient's life (N= 81) | -1.4 (0.8)

21. Secondary Outcome: Caregiver: Degree of Relief of Breakthrough Pain Achieved by Instany at Study End
Description: 0=no reduction, 1=slight, 2=medium, 3=strong, 4=very strong, 5=complete
Time Frame: after therapy with Instanyl (planned: 4 weeks)
Population: Patients included and treated with caregiver documentation (without imputation of missing values), ITT.
  All patients with valid values at last visit. N= number of valid cases (=67). From the 70 participants analyzed, only 67 participants had valid values at the last visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregiver at Final Visit
Number analyzed (Participants) | 70
units on a scale | 3.3 (1.0)

22. Secondary Outcome: Caregiver: Assessment of Breakthrough Pain Therapy by Instanyl (Last Visit)
Description: Scale: 1=very good, 2=good, 3=satisfactory, 4=poor, 5=very poor, 6=insufficient
Time Frame: after therapy with Instanyl (first/last visit)
Population: Patients included and treated with caregiver documentation (without imputation of missing values), intention to treat.
  All patients with valid values ('as observed'). N= number of valid cases.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregiver at Final Visit
Number analyzed (Participants) | 70
units on a scale
  speed of action (N=69) | 2.2 (0.8)
  strength of action (N=69) | 2.1 (0.9)
  tolerability (N=69) | 1.9 (0.8)
  safety (N=68) | 2.0 (0.8)
  handling (N=69) | 2.2 (1.1)
  patient satisfaction (N=68) | 2.1 (1.0)

23. Secondary Outcome: Caregiver: To What Extent Changes Have Occurred Induced by the Treatment of Breakthrough Pain With Instanyl With Respect to ... (at Last Visit)
Description: as for outcome 20
Time Frame: after therapy with Instanyl (at last visit)
Population: Patients included and treated with caregiver documentation (without imputation of missing values), ITT.
  All patients with valid values ('as observed') =N.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregiver at Final Visit
Number analyzed (Participants) | 70
units on a scale
  Nursing and support efforts (N= 69) | -0.8 (0.8)
  Autonomy of the patient (N= 69) | -1.2 (0.8)
  Pain-related impairment in everyday life (N= 69) | -1.3 (0.8)
  Quality of patient's life (N= 68) | -1.3 (0.7)
  Extent of use of other medical services (N= 69) | -0.9 (0.8)

24. Secondary Outcome: Caregiver: To What Extent the Treatment Needs of Your Patient Has Changed by the Use of Instanyl Regarding ...
Description: Scale: -3= very much less, -2= much less, -1= less, 0=comparable, 1= more, 2= much more, 3= very much more
Time Frame: after therapy with Instanyl (last visit)
Population: Patients included and treated with caregiver documentation (without imputation of missing values), ITT.
  All patients with valid values ('as observed'). N= number of valid cases
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregiver at Final Visit
Number analyzed (Participants) | 70
units on a scale
  persistent pain (N=68) | -1.2 (0.9)
  breakthrough pain (N=68) | -1.8 (0.8)
  nausea (N=68) | -1.1 (1.0)
  vomiting (N=65) | -0.9 (1.0)
  dyspnoea (N=66) | -1.1 (1.1)
  constipation (N=68) | -0.8 (1.1)
  weakness (N=68) | -0.7 (0.9)
  poor appetite (N=68) | -0.7 (1.0)
  tiredness (N=67) | -0.8 (1.0)
  efforts due to wounds/decubitus (N=68) | -0.8 (1.0)
  need for assistance in daily activities (N=68) | -1.1 (1.0)
  depressiveness (N=67) | -1.0 (1.1)
  anxiety (N=67) | -1.2 (1.1)
  tension (N=67) | -1.1 (1.0)
  disorientation, confusion (N=67) | -0.9 (1.1)
  Problems with the organization of care (N=68) | -1.0 (1.1)
  Overburdening family/environment (N=68) | -1.2 (1.1)

ADVERSE EVENTS:
Time Frame: First until last visit (planned 4 weeks)
Description: Patients included and treated with at least one application of Instanyl
Arm/Group | All Patients Treated
Serious Adverse Events (participants affected / at risk) | 19/131
Other Adverse Events (participants affected / at risk) | 0/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients Treated (N=131)
Death (General disorders) | 18 (18)
Osteosynthesis (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No